CLINICAL TRIAL: NCT02539433
Title: Imaging of Neuroendocrine Tumors With PET and Fluoro-18-DOPA (F-DOPA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Josephine Rini, Physician, North Shore-LIJ Center for Advanced Medicine, Northwell Health
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: IRB #03-117
Record Dates: First submitted 2015-06-04; First posted 2015-09-03 (Estimated); Last update posted 2015-09-03 (Estimated); Status verified 2015-08

CONDITIONS: Neuroendocrine Tumors
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — fluorodopa F 18

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- F-18-F-DOPA i.v. (Experimental): F-18-F-DOPA i.v. one injection of a dose of up to 8.5 mCi (millicurie). Standard PET scanning started 60-90 minutes post injection.
  Interventions: Procedure: F-18-F-DOPA

INTERVENTIONS:
Procedure: F-18-F-DOPA — F-18-F-DOPA i.v. injection of a dose of up to 8.5 mCi. PET scanning started 60-90 minutes post injection
  Other Names: F-18 fluorodopa

SUMMARY:
Imaging of neuroendocrine (NETs), such as carcinoids and pheochromocytomas (PHEOs), is suboptimal, limiting curative treatment. The investigators wanted to explore the use of PET and F-DOPA i.v. for the localization of these types of neoplasms. The investigators used a similar protocol as they had used for PET (Positron emission tomography) or FDG (Fludeoxyglucose) imaging in oncologic patients. F-DOPA, prepared according to United States Pharmacopeia (USP) guidelines, was approved by the North Shore University Hospital Radiation Safety Committee in 1989 and 1994 for the study of neurological diseases and used uneventfully.

DETAILED DESCRIPTION:
Background: Pre surgical conventional imaging of neuroendocrine tumors (NETs) with CT, MRI, In-111 octreotide or 1-123-MIBG (metaiodobenzylguanidine) scintigraphy has limitations. This pilot study tried to improve the localization of these tumors with F-18-F-DOPA PET scanning.

Methods: The investigators studied 22 patients, the majority referred with clinical diagnosis of carcinoid (9) or NETs (9) and a few with pheochromocytoma/paraganglioma (3). Carbidopa was administered prior to the F-DOPA injection in 12 patients. Comparison was made with prior conventional imaging. The F-DOPA findings, read blindly to the findings of other modalities, were compared with results of subsequent surgery (2), endoscopy (1), or a long-term follow up of mean duration of 49 months (for 20 patients). Two subjects were lost to follow-up.

ELIGIBILITY:
* Inclusion Criteria:

  * 23 years of age and older
  * Appropriate diagnosis by referring physician
* Exclusion Criteria:

  * Less than 23 years of age
  * Greater than 81 years of age
  * Pregnancy
  * Lactation
  * Prior history of radiation treatment
  * Chemotherapy or anti-tuberculosis medications.

Ages: 23 Years to 81 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2003-12; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Imaging of Neuroendocrine Tumors | Mean duration 49 months
  The investigators expect F-18-DOPA to be taken substantially by carcinoid or pheochromocytoma. The outcome for the study is to identify the location of the neoplasm(s) and compare this data with the clinical OctreoScan or I-131 MIBG performed. If the PET/DOPA scan shows different information than the clinical scan that will be communicated to the referring physician. Efforts will be made to collect information regarding the clinical outcome of the patient, further anatomical imaging and/or surgical pathology results.

CONTACTS AND LOCATIONS:
Overall Officials: Josephine Rini, MD, Principal Investigator — North Shore University Hospital
Locations (1):
- North Shore University Hospital, Manhasset, New York, United States

REFERENCES:
- [Result] Neuroendocrinology 2006;83:27-64 DOI: 10.1159/000093339 Published online: May 15, 2006 3rd Annual ENETS Conference March 22-24, 2006, Prague, Czech Republic. Imaging of Neuroendocrine Tumors Zanzi I., Warner R.R.P., Babchyck B., Studentsova Y., Bjelke D., Belakhlef A., Margouleff D., Chaly T. North Shore University Hospital, Manhasset, New York University School of Medicine, New York, N.Y., USA